CLINICAL TRIAL: NCT04920214
Title: Application Value of CEUS Li-RADS in Hepatic Focal Lesions in Patients With Non-high Risk Factors for Hepatocellular Carcinoma
Brief Title: Application Value of CEUS Li-RADS in Hepatic Focal Lesions in Patients With Non-high Risk Factors for HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Tianjin Third Central Hospital (Other); Sichuan Provincial People's Hospital (Other); Fujian Cancer Hospital (Other Government); Jining First People's Hospital (Other); General Hospital of Ningxia Medical University (Other); Beijing Hospital (Other Government); Red Cross Hospital, Hangzhou, China (Other); Zhejiang Cancer Hospital (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1010
Record Dates: First submitted 2021-05-30; First posted 2021-06-09 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver; liver imaging; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: 1. patients with hepatic focal lesions
  2. patients with non-high risk factors for hepatocellular carcinoma
  Interventions: Diagnostic Test: SonoVue

INTERVENTIONS:
Diagnostic Test: SonoVue — CEUS examination was performed and corresponding image information of liver lesions was obtained.

SUMMARY:
Currently, there are few studies on the diagnostic ability of CEUS-LI-RADS in patients with non-high risk factors for liver nodules. Whether this classification is applicable to such patients remains controversial. There are relatively few studies on the diagnostic efficacy of HCC in clinical diagnosis and the consistency between map readers, and the applicable population is only focused on patients with hepatic fibrosis. Therefore, this study explored the application value of CEUS Li-RADS in liver focal lesions in patients with non-high risk factors for hepatocellular carcinoma.

DETAILED DESCRIPTION:
According to the latest epidemiological survey in 2018, primary liver cancer is the sixth most common cancer in the world. Among these, hepatocellular carcinoma is the most common type of liver cancer. Clinicians' diagnosis of HCC has been gradually transformed from invasive puncture diagnosis to non-invasive diagnosis based on enhanced imaging findings. In HCC tissue, the number of small blood vessels was increased and the arrangement was disordered. Compared with the surrounding normal liver tissue, there were more obvious manifestations of increased arterial blood supply. Contrast-enhanced Ultrasound (CEUS) is the most sensitive and objective tool for detecting circulatory perfusion, and can achieve a clear and dynamic display of low speed and small blood flow. Its diagnostic efficacy of HCC is similar to the diagnostic ability of Enhanced CT.

In order to better standardize the writing of liver CEUS report by sonographers, and to facilitate sonographers and clinicians to reach a consensus on the diagnosis and treatment of liver lesions, In 2017, the American Radiology College (ACR) released the CEUS-based Liver Imaging Reporting and Data System (CEUS-Li-RADS). At the same time, according to the perfusion methods in the arterial, portal and venous phases, the CEUS-Li-RADS angiographic findings were classified into main features and LR-M features by ACR Association. The former included high enhancement in arterial phase and mild clearance in portal vein phase (after 60S) or delayed phase. The latter includes annular high enhancement, early clearance and complete clearance. In the classification, CEUS Li-RADS was classified into the following categories according to the possibility of HCC diagnosis with different characteristics of CEUS: LR-1 (definitely benign), LR-2 (possibly benign),LR-3 (possibly HCC), LR-4 (highly suspected HCC), LR-5 (confirmed HCC), and LR-M (liver malignant lesion, not specifically HCC).

In January 2018, Professor Bruix, Chairman of AASLD, wrote in the journal Heaptology that a qualified LIRADS classification should meet the following requirements :(1) LIRADS classification should focus on high-risk groups for HCC; (2) In LI-RADS classification, the specificity of LR-5 in the diagnosis of HCC should be close to 100%; (3) There is a good consistency between the main evaluation criteria of LI-RADS classification, LR-M evaluation criteria and the readers of final classification.

Currently, there are few studies on the diagnostic ability of CEUS-LI-RADS in patients with non-high risk factors for liver nodules. Whether this classification is applicable to such patients remains controversial. There are relatively few studies on the diagnostic efficacy of HCC in clinical diagnosis and the consistency between map readers, and the applicable population is only focused on patients with hepatic fibrosis. Therefore, this study explored the application value of CEUS Li-RADS in liver focal lesions in patients with non-high risk factors for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The patient showed focal liver lesions on routine ultrasound examination.
* Non-HCC high-risk patients (hepatitis B, cirrhosis)

Exclusion Criteria:

* High-risk patients with HCC (hepatitis B, cirrhosis);
* Patients with solid liver tumors could not be found by conventional imaging;
* Patients who do not sign informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. patients with focal liver lesions
  2. patients with non-high risk factors for hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value | 3 years
  The positive predictive value of LR-5 diagnosis of HCC was compared among different map readers
Negative Predictive Value | 3 years
  The negative predictive value of LR-5 diagnosis of HCC was compared among different map readers
Sensitivity | 3 years
  The sensitivity of LR-5 diagnosis of HCC was compared among different map readers
Specificity | 3 years
  The specificity of LR-5 diagnosis of HCC was compared among different map readers

CONTACTS AND LOCATIONS:
Overall Officials: Pintong Huang, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (10):
- China (10):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Shengjing Hospital, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Jining No.1 People's Hospital, Jining, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Red Cross Hospital, Hangzhou, China, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang